CLINICAL TRIAL: NCT06925009
Title: Airway Coach Project: Prediction of Videolaryngoscopy Strategy With Clinical and Ultrasound Parameters (Unicentric)
Status: Recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: MAFV 1
Record Dates: First submitted 2025-03-11; First posted 2025-04-13 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-01

CONDITIONS: Difficult Videolaryngoscopy
Keywords: Ultrasound;Difficult Videolaryngoscopy; Machine Learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient undergoing general anesthesia with videolaryngoscopy intubation: Patient undergoing general anesthesia with intubation We will explore clinical airway parameters and external ultrasound parameters of the airway.
  Interventions: Diagnostic Test: Ultrasound mesurements

INTERVENTIONS:
Diagnostic Test: Ultrasound mesurements — Compare various clinical test with ultrasound parameters to predict difficult videolaryngoscopy intubation.

SUMMARY:
This unicentric observational study collects clinical characteristics, demographic data, and point-of-care airway ultrasound measurements in patients undergoing videolaryngoscopy. These variables are analysed using machine-learning techniques to examine their association with predefined videolaryngoscopy-related outcomes, including blade performance and adjunct requirement.

DETAILED DESCRIPTION:
Tracheal intubation is a routine procedure in anaesthesia and critical care; however, difficulties during videolaryngoscopy may still occur despite advances in airway devices. Conventional bedside airway assessments provide limited guidance for videolaryngoscopy-specific decisions, such as blade selection or anticipation of adjunct use.

This unicentric observational study collects clinical characteristics, demographic data, and point-of-care airway ultrasound measurements in patients undergoing videolaryngoscopy. These variables are analysed using machine-learning techniques to examine their association with predefined videolaryngoscopy-related outcomes, including blade performance and adjunct requirement.

The primary objective is to develop and internally evaluate a predictive model integrating multimodal data to support videolaryngoscopy strategy planning. The model is intended solely as a research and decision-support tool and does not replace clinician judgement. External validation in independent cohorts is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) ASA I-III, aged between 18 and 90 years, undergoing scheduled surgery requiring orotracheal intubation. The signature of the informed consent is required authorizing its inclusion in the study.

Exclusion Criteria:

* Obesity class II defined as a BMI greater than 35.
* Pregnant.
* Cervical tumors, goiter or patients who have required radiotherapy at the cervical level
* Abnormalities that condition anatomy alterations such as facial / cervical fractures.
* Maxillofacial abnormalities
* People who cannot give their consent

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (male or female) ASA I-III, aged between 18 and 90 years, undergoing scheduled surgery requiring orotracheal intubation. The signature of the informed consent is required authorizing its inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Distance from skin to Hyoid bone measured with lineal ultrasound probe | 5 minutes
Distance from skin to epiglottis measured with lineal ultrasound probe | 5 minutes
Tongue Thickness measured with convex probe | 5 minutes
Distance from Jaw to Hyoid bone distance measured with convex probe | 5 minutes

SECONDARY OUTCOMES:
Modified Mallampati Score Class I: Soft palate, uvula, fauces, pillars visible. Class II: Soft palate, major part of uvula, fauces visible. Class III: Soft palate, base of uvula visible. Class IV: Only hard palate visible. | 1minute
Thyromental distance measured from the thyroid notch to the tip of the jaw with the head extended | 1minute
Sternomental distance the distance from the suprasternal notch to the mentum and is measured with the head fully extended on the neck and the mouth closed | 1minute
Interincisor distance DIstance in centimeters between fornt incisors | 1minute
Upper Lip Bite Test upper lip bite criteria-class I = lower incisors can bite the upper lip above the vermilion line, class II = lower incisors can bite the upper lip below the vermilion line, and class III = lower incisors cannot bite the upper lip | 1minute
neck circumference Using a flexible measuring tape in centimeters, neck circumference at the level of thethyroid cartilage will be measured | 1minute

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Universidad de Navarra, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided